CLINICAL TRIAL: NCT02828995
Title: Evaluating the Influence of Diabetes Stigma on Medication Adherence
Acronym: ENDSTIGMA
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Kerri Cavanaugh, Associate Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: 160986
Record Dates: First submitted 2016-06-20; First posted 2016-07-12 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Stigma; Social Determinants of Health
MeSH Terms: conditions — Diabetes Mellitus; Social Stigma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Comprehensive Diabetes Stigma Survey: Participants in the END STIGMA study will be adult patients who have been receiving diabetes-related medical care for a minimum of 12 months in the Vanderbilt University Medical Center Diabetes Clinic and who take at least 1 medication to manage their diabetes.
  Interventions: Other: Comprehensive Diabetes Stigma Survey

INTERVENTIONS:
Other: Comprehensive Diabetes Stigma Survey — The surveys to be administered in the ENDSTIGMA study are as follows:
  1. The Adherence to Refills and Medications for Diabetes survey is a validated, diabetes-specific survey measure utilizing patient self-report to assess diabetes medication adherence.
  2. The Demographics survey will be used to assess participant baseline characteristics, including body mass index (BMI). The questions contained in this survey have been validated by Dr. Kerri Cavanaugh's research group.
  3. Comprehensive Diabetes Stigma Survey is a novel survey being developed and validated in the ENDSTIGMA study. The ENDSTIGMA study will also compare the results from this survey with the medication adherence results, to determine if there is an association between diabetes stigma and medication adherence.

SUMMARY:
The "Evaluating the iNfluence of Diabetes STIGma on Medication Adherence: The ENDSTIGMA Study" was designed to develop a comprehensive diabetes stigma survey measure. The draft measure will be piloted with approximately 50 patients visiting the Vanderbilt University Medical Center (VUMC) Diabetes Clinic. This pilot data will be used to validate the new survey measure and to determine if any questions in the diabetes stigma measure are predictive of diabetes medication adherence.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a chronic condition affecting an estimated 422 million adults worldwide and 28.9 million adults in the US. DM can lead to increased risk of mortality and significant complications including amputation, blindness, cardiovascular disease, and kidney damage. The risk of developing these outcomes can be mediated by early diagnosis and treatment, such as by patient self-management by lifestyle changes and/or taking medication. However, outcome improvement depends on control of blood glucose levels, which in turn depend on adherence to treatment. Several psychosocial factors are known to affect treatment adherence for chronic conditions, one of which is stigma.

Stigma arises when social norms result in the marginalization of people with a certain identity or trait. Negative stereotypes of people in the stigmatized group result in their systematic exclusion and/or discrimination. Chronic disease diagnosis itself can lead to the development of disease-specific identity-based stigma, in that a person's identity is disrupted by a new label (e.g. "diabetic") applied to them, until they incorporate this new label into a positive sense of self. Minority stress theory describes the impact of identity-based marginalization on health outcomes. According to minority stress theory, discrimination and stigma may lead to heightened stress levels, which can translate over time into heightened mental and physical health disparities for the stigmatized group. Categories of stigma experienced by patients include enacted stigma, perceived stigma, self-stigma, and concealment. Enacted stigma refers to acts of discrimination against people in a stigmatized group. Perceived stigma refers both to the fear of experiencing enacted stigma, as well as to the shame resulting from belonging to or being associated with a stigmatized group. Self-stigma refers to the internalization of negative group stereotypes by members of the stigmatized group. Concealment, also called non-disclosure, refers to the hiding of a stigmatized identity or condition.

Stigma has been shown to negatively affect access to care as well as quality of life in people living with chronic diseases. Disease-specific stigma scales have been developed for various conditions, including mental illness, HIV/AIDS, epilepsy, and obesity. These scales have been used to facilitate interventions to minimize negative effects of stigma on health behaviors and outcomes. In comparison to other health conditions, diabetes stigma has only recently emerged as a research topic of interest.

DM has been reported to be a health condition that is relatively less stigmatized in comparison to other conditions. One publication suggested in its introduction that "diabetes does not appear to have associated stigma." As such, there have been publications comparing the degree of stigma experienced by DM patients with those with conditions such as schizophrenia, dementia, HIV, depression, and hypertension. However, numerous qualitative studies interviewing people with diabetes have revealed that DM patients do experience significant disease-related stigma.

In the literature, DM-related enacted stigma examples include workplace discrimination (decreased chance of being hired and increased chance of job loss); threatened or actual termination of romantic relationships; and judgmental behavior from healthcare professionals. Likewise, examples of perceived stigma include fear of being characterized as an illicit drug user when injecting insulin in public; and feelings of isolation when choosing to eat different foods, particularly in family and cultural situations. Self-stigma and concealment examples include avoidance of social events; timing self-management so it can be done in isolation; and altering blood glucose recordings, so as to appear "healthy."

Despite ample evidence of the existence of DM-specific stigma, limited attempts have been made to measure it. The Diabetes Distress Scale (DDS) was designed to measure "emotional burden, physician-related distress, regimen-related distress, and…interpersonal distress" associated with DM. However, the DDS does not comprehensively measure all the types of stigma minority stress theory has shown to contribute to chronic disease health disparities. The Barriers to Diabetes Adherence measure includes six questions about stigma, but the scope of these questions was limited and targeted towards an adolescent population with Type 1 DM. A limited number of previous publications have adapted disease-specific stigma scales from other conditions or developed their own questionnaires for said conditions for their diabetes stigma research needs. To date, only one publication has developed and validated a stigma scale specifically for DM patients, and this measure only addressed self-stigma. Therefore, to our knowledge, there is currently no scale that measures multiple facets of DM-specific stigma that may be contributing to sub-optimal patient diabetes self-management. Given the relationship between stigma, treatment adherence, and adverse health outcomes for chronic disease patients, development of a comprehensive DM stigma scale may lead to improvements in DM patient centered care, which will be addressed by the following Specific Aims:

Specific Aims

1. Develop a novel quantitative measure that comprehensively measures enacted stigma, perceived stigma, and self-stigma and concealment specific to adult DM patients
2. Pilot the measure with 30-50 DM patients
3. Validate the measure and determine if DM stigma is associated with obesity, diabetes type, insulin use, and/or is predictive of medication adherence

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Type I or II DM for at least 1 year
* Taking at least 1 medication to manage diabetes

Exclusion Criteria:

* Under 18 years of age
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be adult patients with an established diagnosis of diabetes and who are taking at least 1 medication to manage their diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Diabetes Stigma | Baseline
  The composite stigma score from the Comprehensive Diabetes Stigma Survey measure will be calculated from patient survey responses.
Diabetes Medication Adherence | Baseline
  The composite diabetes medication adherence score will be calculated from patient responses to the Adherence to Refills and Medications Scale - Diabetes (ARMS-D) survey.

SECONDARY OUTCOMES:
Diabetes Patient Height (in Inches) | Baseline
  Self-Report of Diabetes Patient Height
Diabetes Patient Weight (in Pounds) | Baseline
  Self-Report of Diabetes Patient Weight

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Cavanaugh, MD/MHS, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. Global report on diabetes. Geneva: World Health Organization, 2016.
- [Background] Centers for Disease Control and Prevention. National Diabetes Statistics Report: Estimates of Diabetes and Its Burden in the United States, 2014. Atlanta: U.S. Department of Health and Human Services, 2014.
- [Background] Stolar M. Glycemic control and complications in type 2 diabetes mellitus. Am J Med. 2010 Mar;123(3 Suppl):S3-11. doi: 10.1016/j.amjmed.2009.12.004. PMID 20206730
- [Background] Egede LE, Gebregziabher M, Echols C, Lynch CP. Longitudinal effects of medication nonadherence on glycemic control. Ann Pharmacother. 2014 May;48(5):562-70. doi: 10.1177/1060028014526362. Epub 2014 Feb 28. PMID 24586059
- [Background] Kato A, Fujimaki Y, Fujimori S, Isogawa A, Onishi Y, Suzuki R, Yamauchi T, Ueki K, Kadowaki T, Hashimoto H. Association between self-stigma and self-care behaviors in patients with type 2 diabetes: a cross-sectional study. BMJ Open Diabetes Res Care. 2016 Jan 5;4(1):e000156. doi: 10.1136/bmjdrc-2015-000156. eCollection 2016. PMID 26835138
- [Background] Link BG, Phelan JC. Conceptualizing stigma. Annu Rev Sociol. 2001;27:363-85.
- [Background] Laws MB. Explanatory Models and Illness Experience of People Living with HIV. AIDS Behav. 2016 Sep;20(9):2119-29. doi: 10.1007/s10461-016-1358-1. PMID 26971285
- [Background] Goldman JB, Maclean HM. The significance of identity in the adjustment to diabetes among insulin users. Diabetes Educ. 1998 Nov-Dec;24(6):741-8. doi: 10.1177/014572179802400610. PMID 10025297
- [Background] Abdoli S, Ashktorab T, Ahmadi F, Parvizy S, Dunning T. Seeking new identity through the empowerment process. Iran J Nurs Midwifery Res. 2014 Mar;19(2):145-51. PMID 24834083
- [Background] Mirowsky J, Ross CE. Social Causes of Psychological Distress. NY: Aldine de Gruyter; 1989.
- [Background] Meyer IH. Prejudice, social stress, and mental health in lesbian, gay, and bisexual populations: conceptual issues and research evidence. Psychol Bull. 2003 Sep;129(5):674-697. doi: 10.1037/0033-2909.129.5.674. PMID 12956539
- [Background] Pearlin LI. The sociological study of stress. J Health Soc Behav. 1989 Sep;30(3):241-56. PMID 2674272
- [Background] Lick DJ, Durso LE, Johnson KL. Minority Stress and Physical Health Among Sexual Minorities. Perspect Psychol Sci. 2013 Sep;8(5):521-48. doi: 10.1177/1745691613497965. PMID 26173210
- [Background] Scambler G, Hopkins A. Being epileptic: Coming to terms with stigma. Sociol Health Illn. 1986;8:26-43.
- [Background] Corrigan PW, Watson AC. The paradox of self-stigma and mental illness. Clin Psychol. 2002;9:35-53
- [Background] Joachim G, Acorn S. Stigma of visible and invisible chronic conditions. J Adv Nurs. 2000 Jul;32(1):243-8. doi: 10.1046/j.1365-2648.2000.01466.x. PMID 10886457
- [Background] Earnshaw VA, Quinn DM. The impact of stigma in healthcare on people living with chronic illnesses. J Health Psychol. 2012 Mar;17(2):157-68. doi: 10.1177/1359105311414952. Epub 2011 Jul 28. PMID 21799078
- [Background] Boyd JE, Adler EP, Otilingam PG, Peters T. Internalized Stigma of Mental Illness (ISMI) scale: a multinational review. Compr Psychiatry. 2014 Jan;55(1):221-31. doi: 10.1016/j.comppsych.2013.06.005. Epub 2013 Sep 21. PMID 24060237
- [Background] Berger BE, Ferrans CE, Lashley FR. Measuring stigma in people with HIV: psychometric assessment of the HIV stigma scale. Res Nurs Health. 2001 Dec;24(6):518-29. doi: 10.1002/nur.10011. PMID 11746080
- [Background] Fernandes PT, Salgado PC, Noronha AL, Sander JW, Li LM. Stigma Scale of Epilepsy: validation process. Arq Neuropsiquiatr. 2007 Jun;65 Suppl 1:35-42. doi: 10.1590/s0004-282x2007001000006. PMID 17581666
- [Background] Lillis J, Luoma JB, Levin ME, Hayes SC. Measuring weight self-stigma: the weight self-stigma questionnaire. Obesity (Silver Spring). 2010 May;18(5):971-6. doi: 10.1038/oby.2009.353. Epub 2009 Oct 15. PMID 19834462
- [Background] Schabert J, Browne JL, Mosely K, Speight J. Social stigma in diabetes : a framework to understand a growing problem for an increasing epidemic. Patient. 2013;6(1):1-10. doi: 10.1007/s40271-012-0001-0. PMID 23322536
- [Background] Fernandes PT, Salgado PC, Noronha AL, Barbosa FD, Souza EA, Sander JW, Li LM. Prejudice towards chronic diseases: comparison among epilepsy, AIDS and diabetes. Seizure. 2007 Jun;16(4):320-3. doi: 10.1016/j.seizure.2007.01.008. Epub 2007 Feb 22. PMID 17320420
- [Background] Lee S, Lee MT, Chiu MY, Kleinman A. Experience of social stigma by people with schizophrenia in Hong Kong. Br J Psychiatry. 2005 Feb;186:153-7. doi: 10.1192/bjp.186.2.153. PMID 15684240
- [Background] Woo BK, Mehta P. Examining the differences in the stigma of dementia and diabetes among Chinese Americans. Geriatr Gerontol Int. 2017 May;17(5):760-764. doi: 10.1111/ggi.12782. Epub 2016 May 2. PMID 27137751
- [Background] Roeloffs C, Sherbourne C, Unutzer J, Fink A, Tang L, Wells KB. Stigma and depression among primary care patients. Gen Hosp Psychiatry. 2003 Sep-Oct;25(5):311-5. doi: 10.1016/s0163-8343(03)00066-5. PMID 12972221
- [Background] Browne JL, Ventura A, Mosely K, Speight J. 'I'm not a druggie, I'm just a diabetic': a qualitative study of stigma from the perspective of adults with type 1 diabetes. BMJ Open. 2014 Jul 23;4(7):e005625. doi: 10.1136/bmjopen-2014-005625. PMID 25056982
- [Background] Browne JL, Ventura A, Mosely K, Speight J. 'I call it the blame and shame disease': a qualitative study about perceptions of social stigma surrounding type 2 diabetes. BMJ Open. 2013 Nov 18;3(11):e003384. doi: 10.1136/bmjopen-2013-003384. PMID 24247325
- [Background] Tak-Ying Shiu A, Kwan JJ, Wong RY. Social stigma as a barrier to diabetes self-management: implications for multi-level interventions. J Clin Nurs. 2003 Jan;12(1):149-50. doi: 10.1046/j.1365-2702.2003.00735.x. No abstract available. PMID 12519263
- [Background] Nebiker-Pedrotti PM, Keller U, Iselin HU, Ruiz J, Parli K, Caplazi A, Puder JJ. Perceived discrimination against diabetics in the workplace and in work-related insurances in Switzerland. Swiss Med Wkly. 2009 Feb 21;139(7-8):103-9. doi: 10.4414/smw.2009.12432. PMID 19234878
- [Background] Hopper S. Diabetes as a stigmatized condition: the case of low-income clinic patients in the United States. Soc Sci Med Med Anthropol. 1981 Jan;15B(1):11-9. doi: 10.1016/0160-7987(81)90004-1. No abstract available. PMID 7209601
- [Background] Kumar K, Greenfield S, Raza K, Gill P, Stack R. Understanding adherence-related beliefs about medicine amongst patients of South Asian origin with diabetes and cardiovascular disease patients: a qualitative synthesis. BMC Endocr Disord. 2016 May 26;16(1):24. doi: 10.1186/s12902-016-0103-0. PMID 27230479
- [Background] Broom D, Whittaker A. Controlling diabetes, controlling diabetics: moral language in the management of diabetes type 2. Soc Sci Med. 2004 Jun;58(11):2371-82. doi: 10.1016/j.socscimed.2003.09.002. PMID 15047092
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Mulvaney SA, Hood KK, Schlundt DG, Osborn CY, Johnson KB, Rothman RL, Wallston KA. Development and initial validation of the barriers to diabetes adherence measure for adolescents. Diabetes Res Clin Pract. 2011 Oct;94(1):77-83. doi: 10.1016/j.diabres.2011.06.010. Epub 2011 Jul 7. PMID 21737172
- [Background] Kato A, Takada M, Hashimoto H. Reliability and validity of the Japanese version of the self-stigma scale in patients with type 2 diabetes. Health Qual Life Outcomes. 2014 Dec 12;12:179. doi: 10.1186/s12955-014-0179-z. PMID 25495723
- [Background] Borson S, Scanlan J, Brush M, Vitaliano P, Dokmak A. The mini-cog: a cognitive 'vital signs' measure for dementia screening in multi-lingual elderly. Int J Geriatr Psychiatry. 2000 Nov;15(11):1021-7. doi: 10.1002/1099-1166(200011)15:113.0.co;2-6. PMID 11113982
- [Background] Mayberry LS, Gonzalez JS, Wallston KA, Kripalani S, Osborn CY. The ARMS-D out performs the SDSCA, but both are reliable, valid, and predict glycemic control. Diabetes Res Clin Pract. 2013 Nov;102(2):96-104. doi: 10.1016/j.diabres.2013.09.010. Epub 2013 Sep 26. PMID 24209600
- [Background] Nam S, Chesla C, Stotts NA, Kroon L, Janson SL. Barriers to diabetes management: patient and provider factors. Diabetes Res Clin Pract. 2011 Jul;93(1):1-9. doi: 10.1016/j.diabres.2011.02.002. Epub 2011 Mar 5. PMID 21382643